CLINICAL TRIAL: NCT00386841
Title: Associations Between Gene-Polymorphisms, Endo-Phenotypes for Depression and Antidepressive Treatment (AGENDA)
Brief Title: Outcome Following Antidepressant Treatment on Possible Endo-Phenotypes for Major Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Lars Vedel Kessing and Ulrik Gether, professors, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: AGENDA
Record Dates: First submitted 2006-10-11; First posted 2006-10-12 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Healthy
Keywords: Major depression; First degree relatives; Escitalopram; Cortisol; Cognition; Personality; Endo-phenotype
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram; Dexetimide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A Escitalopram 10 mg (Active Comparator): Escitalopram 10 mg
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram — Escitalopram 10 mg p.o. per day
  Other Names: cipralex
  Arms: A Escitalopram 10 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether outcome following antidepressant treatment can be used as a tool to evaluate endo-phenotypes for depression.

DETAILED DESCRIPTION:
The research in depression has for some years focused at the identification of endo-phenotypes. Endo-phenotypes are heritable biological or psychological markers, which are more commonly found in patients and their healthy relatives than in the general population.

Recent studies point at disturbed regulation of the hypothalamic-pituitary-adrenocortical (HPA) system as a possible endo-phenotype for depression.

The hypothesis of AGENDA are that endo-phenotypes are affected by treatment with antidepressants in healthy first degree relatives.

AGENDA is a four week randomized, placebo-controlled, double-blind trial in which first degree relatives of patients with the diagnosis of depression are randomised in to two groups, which are treated with either placebo or antidepressant medicine (Cipralex). We expect to include 80 healthy subjects, with the predisposition for depression, since one of their parents or siblings recently was treated for depression.

The subjects will be examined before and after four weeks of treatment by a thorough interview concerning psychiatric symptoms (SCAN), including depressive symptoms, personality, perceived stress and cognitive function. The effect of antidepressant on stress is measured with saliva-cortisol and by the response to the combined dexamethasone corticotropin-releasing (CRH) hormone test. Additionally, MR and PET scans of the 5-HT4 receptor function will be conducted before and after 4 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Offsprings or siblings of patients with major depression
* Born in Denmark with European parents and grandparents
* For women; not pregnant or breastfeeding
* Written informed consent

Exclusion Criteria:

* Somatically illness or other handicaps which make participation in the study impossible
* Daily intake of drugs interfering with corticosteroids or escitalopram
* Hypersensitivity to escitalopram, dexamethasone or human corticotropin-releasing hormone
* Former medical or psychological treatment for diseases in the affective or schizophrenic spectrum
* Ongoing addiction of alcohol or psychoactive drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2007-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Changes in the response on the combined dexamethasone corticotropin-releasing hormone test before and after 4 weeks treatment with escitalopram or placebo. | 4-6 weeks

SECONDARY OUTCOMES:
Changes in scores before and after 4 weeks treatment with escitalopram or placebo on: Cognition | 4-6 weeks
Social function | 4-6 weeks
Neuroticism | 4-6 weeks
Subjective; sleep, pain, aggression, depression, anxiety, quality of life, perceived stress and side-effects | 4-6 weeks
Receptor status by PET-scans | 4-6 weeks
Inflammatory parameters | 4-6 weeks
Paraclinical measures | 4-6 weeks
MR and fMRI | 4-6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lars V Kessing, DMSc, Study Director — Psychiatric Department of Rigshospitalet, Blegdamsvej 9, DK-2100 Copenhagen OE
Locations (1):
- Psychiatric Department of Rigshospitalet, Blegdamsvej 9, Copenhagen OE, Denmark

REFERENCES:
- [Derived] Knorr U, Vinberg M, Mortensen EL, Winkel P, Gluud C, Wetterslev J, Gether U, Kessing LV. Effect of chronic escitalopram versus placebo on personality traits in healthy first-degree relatives of patients with depression: a randomized trial. PLoS One. 2012;7(2):e31980. doi: 10.1371/journal.pone.0031980. Epub 2012 Feb 29. PMID 22393376
- [Derived] Knorr U, Vinberg M, Hansen A, Klose M, Feldt-Rasmussen U, Hilsted L, Hasselstrom J, Gether U, Winkel P, Gluud C, Wetterslev J, Kessing LV. Escitalopram and neuroendocrine response in healthy first-degree relatives to depressed patients--a randomized placebo-controlled trial. PLoS One. 2011;6(6):e21224. doi: 10.1371/journal.pone.0021224. Epub 2011 Jun 27. PMID 21738622
- [Derived] Knorr U, Vinberg M, Klose M, Feldt-Rasmussen U, Hilsted L, Gade A, Haastrup E, Paulson O, Wetterslev J, Gluud C, Gether U, Kessing L. Rationale and design of the participant, investigator, observer, and data-analyst-blinded randomized AGENDA trial on associations between gene-polymorphisms, endophenotypes for depression and antidepressive intervention: the effect of escitalopram versus placebo on the combined dexamethasone-corticotrophine releasing hormone test and other potential endophenotypes in healthy first-degree relatives of persons with depression. Trials. 2009 Aug 11;10:66. doi: 10.1186/1745-6215-10-66. PMID 19671139